CLINICAL TRIAL: NCT05613699
Title: Implementation and Evaluation of Physical Exercise Services for Young Adults With Cancer
Brief Title: Exercise for Young Adults With Cancer
Acronym: YOUEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Charite University, Berlin, Germany (Other); University Clinic Cologne (Unknown); University Clinic Essen (Unknown)
Responsible Party: Principal Investigator, Joachim Wiskemann, Head Exercise Oncology, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YOUEX_S932
Record Dates: First submitted 2022-10-17; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Fatigue; Cancer; Physical Activity; Exercise
Keywords: cancer; social media; exercise; virtual training; app
MeSH Terms: conditions — Fatigue; Neoplasms; Motor Activity; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- supervised, group-based, online-social media exercise program (Other)
  Interventions: Behavioral: Exercise - Social Media
- unsupervised individual home-based training with an online-training app (Other)
  Interventions: Behavioral: Exercise - App
- supervised, in-person exercise program close to place of residence (Other)
  Interventions: Behavioral: Exercise - closed to patients residence

INTERVENTIONS:
Behavioral: Exercise - Social Media — The supervised online-social media exercise intervention took place once per week at a fixed, pre-scheduled time, via an online video conference platform. The training sessions lasted for 60 minutes and included a holistic workout with different focuses (e.g. resistance training for lower extremities, sensorimotor training, home-based endurance training). Patients were further recommended independent physical activity like walking or cycling, 1-2 times per week or to maintain the current volume of physical activity.
  Arms: supervised, group-based, online-social media exercise program
Behavioral: Exercise - App — Exercise program in the online-app were personalized and focused on a combination of endurance and resistance training, 2-3 times a week, depending on patient's needs. Additional types of exercise (e.g. sensorimotor training) were added if therapy-related side effects were present. If necessary, exercise trainers conducted one introductory training session as video conference to check for exercise techniques and answer any individual questions.
  Arms: unsupervised individual home-based training with an online-training app
Behavioral: Exercise - closed to patients residence — The supervised exercise program close to patient's home was executed in a certified exercise facility of the network OnkoAktiv and supervised by special qualified exercise trainers. The weekly recommendation was to participate in a personalized in-person exercise program 1-2 per week, plus independent physical activity (or to maintain current level of physical activity)
  Arms: supervised, in-person exercise program close to place of residence

SUMMARY:
Over the past decade, importance of supportive care in cancer treatment of young cancer patients has increased. However, most common cancer-related side effects, such as physical deconditioning, psychological problems, infertility, and cancer-related fatigue, are particularly problematic for young adults (AYA). Short- and long-term side effects result in impaired quality of life, social life, and physical activity levels. While there is growing evidence that physical exercise is effective in reducing disease- or treatment-related side effects, programs are generally not tailored to the unique needs of young adults. In addition, social media or web-based programs are rarely structurally integrated into existing care programs. The objective of the Your Exercise Program (YOUEX) study is therefore to address these specific needs and to improve physical exercise services for young people in Germany. To this end, this pilot study presents three approaches to physical activity enhancement, with a particular focus on web-based and cross-regional programs. All three approaches will be evaluated for their feasibility and effectiveness on fatigue, distress, quality of life, and activity levels, as well as sustained effects over 24 weeks. The YOUEX study is an exploratory intervention study in the form of a 12-week exercise program for patients aged 18 to 39 years who currently have or have had a cancer diagnosis within the past 5 years. Eligible patients can choose from three support programs: Social Media Exercise Program, Online Exercise Platform, Supervised Exercise Program. The goal is to recruit 70 to 80 patients over an 8-month period. Evaluation questionnaires will be sent at three time points (T0: start of exercise program, T1: after 6 weeks; T2: after 12 weeks; T3: after 24 weeks) with a short weekly questionnaire between T0 and T2 to assess weekly adherence and changes in fatigue. YOUEX study will collect detailed information on the acceptability and feasibility of different physical activity programs for young people and their lasting effects on fatigue, quality of life and physical activity. Should these be positive, the findings can directly inform health care practice, which would be highly relevant especially in light of the COVID pandemic.

ELIGIBILITY:
Inclusion Criteria:

* cancer diagnosis within the past five years
* signed informed consent

Exclusion Criteria:

* cancer-related cognitive impairment
* lack of sports clearance from the attending oncologist (e.g. in case of fragile bone metastases)
* current participation in another exercise intervention
* insufficient German language skills

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the three exercise interventions | During 12 week of the intervention
  Participants ability to follow the exercise prescription (measured by % of training frequency as well as type of the exercise)

SECONDARY OUTCOMES:
Physical activity level | 12 weeks and 24 weeks
  Physical activity levels were determined by the standardized Godin-Shephard Leisure-Time Questionnaire. The questionnaire was used to ask for pre-diagnosis-, post-diagnosis- and pre-post-intervention physical activity levels within three categories: light, moderate and vigorous physical activity in minutes per week. Participants were categorized in an active and inactive subgroup with a threshold of 150 minutes moderate or 75 minutes vigorous physical activity per week (or the combination of both) based on the American College of Sports Medicine (ACSM) guidelines.
Module Selection and preferences | Baseline, 6 weeks, 12 weeks
  The individual module selection and preferences were queried and documented at the first three time points (Baseline, after 6 week and after 12 weeks). Reasons for any module selection and why other modules have not been selected were collected through open answer questions while multiple answers were possible. The subgroups of the initial module selection were analyzed according treatment and employment status. Further, we asked for module preferences under COVID-19 free conditions
Impact of COVID-19 pandemic | Baseline, 6 weeks, 12 weeks, 24 weeks
  The questionnaire about the impact of COVID-19 has been self-developed, but internal validated in other studies at the National Center of Tumor Diseases (NCT) Heidelberg. The COVID-19 questionnaire consisted of six items and surveyed the impact of COVID-19 on patient´s current job situation, leisure-time activities, physical activity levels, self-efficacy, anxiety and mental health. Further we asked for, whether COVID-19 had any effect on the participants module selection. The COVID-19 questionnaire was submitted later during the ongoing study due to COVID-19-lockdown in November 2020. Therefore, not all participants completed the COVID-19 questionnaire
Fatigue | Baseline, 6 weeks, 12 weeks, 24 weeks
  Standardized questionnaire used: European Organisation for Research and Treatment of Cancer (EORTC) FA (Fatigue) 12
Health-related quality of life | Baseline, 6 weeks, 12 weeks, 24 weeks
  Quality of life (QoL) will be assessed with the validated 30-item self-assessment questionnaire of the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0). It includes five multi-item functional scales (physical, role, emotional, cognitive, and social function), three multi-item symptom scales (fatigue, pain, nausea/vomiting), and six single items assessing further symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea) and financial difficulties.
Distress | Baseline, 6 weeks, 12 weeks, 24 weeks
  Standardized questionnaire used: National Comprehensive Cancer Network (NCCN) Distress-Thermometer
Patient Satisfaction | Baseline, 6 weeks, 12 weeks, 24 weeks
  Standardized questionnaire used: Zufriedenheit (ZUF)-8 Questionnaire
Social Support | Baseline, 6 weeks, 12 weeks, 24 weeks
  Standardized questionnaire used: German translation of the questionnaire by Sallis (1987)
Fatigue Thermometer | Daily till week 12
  Standardized questionnaire used: Style of NCCN Distress-Thermometer. Dimensions: Physical, emotional and mental Fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wiskemann, PhD, Principal Investigator — Heidelberg University Hospital / National Center for Tumor Diseases
Locations (1):
- National Center for Tumor Diseases, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Voland A, Krell V, Gotte M, Niels T, Koppel M, Wiskemann J. Exercise Preferences in Young Adults with Cancer-The YOUEX Study. Curr Oncol. 2023 Jan 21;30(2):1473-1487. doi: 10.3390/curroncol30020113. PMID 36826074